CLINICAL TRIAL: NCT03644849
Title: A Single Center, Prospective, Double-blinded, Randomized, Placebo-controlled Trial Evaluating the Efficacy of Fractionated Carbon Dioxide Therapy in Postoperative Lower Extremity Wound Healing
Brief Title: Evaluating the Safety and Efficacy of Fractionated Carbon Dioxide Therapy in Postoperative Lower Extremity Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Ramona Behshad, MD, Assistant Professor Department of Dermatology, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 29076
Record Dates: First submitted 2018-08-13; First posted 2018-08-23 (Actual); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Leg Ulcer
Keywords: Leg Ulcer; Lower extremity ulcer; carbon dioxide laser; CO2 Laser; Ablative fractional carbon dioxide lasers
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Fractional carbon dioxide laser intervention group (Experimental): The intervention will only involve a single treatment with ablative fractional carbon dioxide laser therapy. The investigators will specifically be using the CO2RE® (Syneron Candela Corp, Wayland, MA).
  Interventions: Device: CO2RE® (Syneron Candela Corp, Wayland, MA)
- Sham laser intervention group (Sham Comparator)
  Interventions: Other: Sham laser treatment

INTERVENTIONS:
Device: CO2RE® (Syneron Candela Corp, Wayland, MA) — The intervention will include a single treatment of a lower extremity wound with ablative fractional carbon dioxide laser after MMS surgery.
  Other Names: Ablative fractional carbon dioxide laser
  Arms: Fractional carbon dioxide laser intervention group
Other: Sham laser treatment — A physician who is not blinded will perform a sham laser treatment on blinded subjects.
  Arms: Sham laser intervention group

SUMMARY:
This study will evaluate the efficacy and safety of laser therapy on postoperative lower extremity wound healing over 12 weeks. The investigators will include adult patients who have underwent Mohs Micrographic Surgery on their lower extremities. Patients with poor immune systems, current pregnancies, uncontrolled diabetes, lower extremity venous or arterial disease will not be included in this study. After surgery patients will be randomized into two groups. One group will receive a single laser treatment immediately after their surgery on their wound while the other will not. The group not receiving laser therapy will undergo a sham laser therapy treatment. Immediately after therapy and 4, 8, and 12 weeks postoperative patients will have a follow up visit. During these visits patients wound size will be recorded, a photograph will be taken, and the wound temperature will be measured. Patient will be given a diary to record any adverse events related to the wound.

DETAILED DESCRIPTION:
Background and Significance

With an aging population, the prevalence of cutaneous malignancies continues to pose significant burden in terms of morbidity and economic cost. It is estimated that 5.4 million new cases of non-melanoma skin cancers, i.e squamous cell carcinoma (SCC) and basal cell carcinoma (BCC), are diagnosed each year. As the incidence of skin cancer increases, the prevalence of postoperative lower extremity wounds also increases. Epidemiologic studies consistently find up to 10% of BCC and 20% of SCC occur on the lower extremity in both men and women, and the largest portion of malignant melanoma cases occurs on the legs of women. Lower extremity ulcers are a common postoperative complication of melanoma, BCC and SCC treatment, and impose an undue health care burden by negatively impacting patient quality of life and increasing costs. Recent reports suggest that lower extremity ulcers cost $10,000 per patient per year, and patients often reported social isolation and depression, thus making an improved treatment protocol for healing lower extremity wounds essential.

After an acute injury, normal wound healing is usually complete within four weeks and can be divided into 4 phases: coagulation, inflammation, formulation of granulation tissue, and remodeling or scar formation. The initial steps of coagulation and inflammation involve the inhibition of bleeding through activation of the coagulation cascade, release of growth factors and cytokines such as platelet-derived growth factor and transforming growth factor β, and recruitment of macrophages and fibroblasts. This facilitates removal of foreign bodies and bacteria while preparing the wound site for new tissue. Around 5-7 days inflammation subsides via apoptosis of proinflammatory cells followed by formation of granulation tissue through dermal and epidermal cell migration to the wound bed. Granulation tissue has a high metabolic demand that is supplied by angiogenesis (proliferation of new blood vessels). Angiogenesis occurs due to local hypoxia during acute tissue injury which stimulates the release of several factors such as vascular endothelial growth factor and fibroblast growth factor 2. Lastly matrix remodeling and scar formation result in the restoration of primarily normal epidermis by replacing the extracellular matrix containing collagen III to primarily collagen I and myofibroblast induced tissue contraction.

Lower extremity ulcers exhibit increased infection risk compared with other body sites, and are rarely amenable to surgical closure due to a lack of suitable local skin and poor tissue vascularity. As a result, many of these defects are allowed to heal via secondary intention healing (SIH).The lower extremity suffers from poor perfusion and hypovascularity, both of which impair wound healing in this anatomic site. Therefore, post-surgical wounds on the lower extremities frequently convert into chronic wounds, defined as wounds that fail to heal within four weeks and show no sign of improvement within eight weeks. This protracted healing course drains the medical system of resources and subjects the patient to significant discomfort and distress. The major problems reported from patients include pain, immobility, sleep disturbances, lack of energy, limitations in work and leisure activities, worry, frustration, and lack of self-esteem. Given the problems associated with allowing lower extremity ulcers to heal by second intent, strategies that improve ulcer healing would be beneficial, improving patient quality of life and preventing further complications.

Ablative fractional carbon dioxide lasers, such as the CO2RE® (Syneron Candela Corp, Wayland, MA), offer a multi-depth pulse technology that delivers a precise fractionated beam pattern to treat the epidermis and dermis simultaneously. This precision technology creates areas of superficial and deep ablation and coagulation to activate remodeling at several tissue depths. The CO2RE® is FDA-approved and has demonstrated efficacy in post-surgical scar treatment, although it has not been studied in acute, lower extremity ulcers.

While the use of AFLs for wounds is novel, there are sufficient reported studies to suggest it may be an efficacious intervention to facilitate the healing of lower extremity surgical wounds. AFLs create microscopic wounds that can reach greater dermal depths than previously attainable with fully ablative devices, and adjacent untreated skin may facilitate rapid healing. Histopathologic studies of normal skin treated with AFL demonstrate altered kinetics of growth factor and cytokine release, expression of heat shock proteins and matrix metalloproteinases. In 3D human organotypic full-thickness skin models, carbon dioxide AF therapy resulted in reduced expression of matrix metalloproteinases, and downregulation of pro-inflammatory cytokines. Therefore, carbon dioxide AFL may offer significant advantages over traditional non-ablative laser technologies.

Mohs Surgery

The treatment for BCC and SCC is often surgical. Mohs Micrographic Surgery (MMS) is a surgical procedure in which skin cancer cells are removed. Once all visibly cancerous tissue is removed, the tissue is examined under a microscope to evaluate for the presence of cancer cells at the tissue edges. This allows the surgeon to determine if all of the cancer has been removed. After examining the specimen, multiple thin sections of tissue are removed around the margins of the wound and then examined under a microscope. If abnormal cells remain, further tissue excision is required. This process is continued until no cancerous cells remain. This technique allows for preservation of maximum amount of normal tissue and the pathologic confirmation of complete cancer excision. MMS is used when there is a high risk of recurrence, when the skin cancer is located in a sensitive area such as the nose or lower extremities, or the cancer is an aggressive subtype. Complications of MMS include infection, hypertrophic scar formation, hypergranulation tissue, and impaired wound healing that can result is ulcers persisting up to 7 months.

Innovation

This project tests the highly innovative hypothesis that use of the AFL is both safe and efficacious for the treatment of post-surgical ulcers. This laser technology has demonstrated efficacy for treatment of lower extremity scars, but has not been adequately evaluated in ulcers. Due to a unique pattern of injury induced by fractional technology where healthy tissue in the vicinity of the ulcer is spared, the use of this technology may demonstrate significant benefits as compared to traditional non-ablative lasers and low level light systems previously used to treat ulcers.

Although our proposed study is highly novel, the feasibility of our proposed protocol is supported by the fact that the fractional carbon dioxide laser has been shown to improve wound healing in scar-related wounds and in post-traumatic wounds of the lower extremity. Based on this data, treating acute lower extremity ulcers with ablative fractional carbon dioxide laser is expected to improve healing times in lower extremity ulcers occurring as a result of cutaneous surgery. This work may lead to the use of ablative fractional laser to support the body's regenerative capacity on the lower extremity, improving patient quality of life and conserving healthcare resources. The investigators therefore hypothesize that ablative fractional laser treatment therapy after cutaneous surgery is a safe and efficacious treatment for lower extremity wounds.

In addition to the novelty of our proposed hypothesis, our study benefits from technical innovation in adjudicating ulcer healing, which has previously not been combined with carbon dioxide laser technology.

Preliminary Studies

The first report of carbon dioxide AFL utilization in wounds was by Schumaker et. al in 2012. In their report they described three patients treated with a 10.6-um carbon dioxide AFL system for multiple traumatic scars related to blast injury. Incidentally they noted that chronic wounds in the treatment sites resolved within 2 weeks of initial therapy. Phillips et. al observed similar results in elderly individuals with post traumatic lower extremity ulcers. Their report demonstrated greater than 60% resolution of chronic lower-extremity ulcers 3 weeks after a single treatment with carbon dioxide AFL therapy. Most recently Krakowski et. al demonstrated near complete resolution of two chronic wounds by two months in pediatric patients after treatment with CO2 AFL at a pulse energy of 50 mJ and treatment density of 5%.

MMS performed on the nose, like lower extremities, are occasionally allowed to heal by second intent and can thus be predisposed to prolonged healing. Our preliminary studies demonstrate the effects of carbon dioxide AFL on these wounds. Two patients receiving MMS on the nasal ala were studied. One patient receiving carbon dioxide AFL therapy on his postoperative wound while the other did not. After three weeks the patient's postoperative wounds were assessed. The patient receiving laser therapy had complete epithelialization of his wound, while the patient with no treatment had incomplete epithelization. These results suggest the hypothesis that the carbon dioxide AFL may be a safe, efficacious treatment for ulcers of the lower extremity.

Design:

Our study is a prospective, double-blinded, randomized, placebo-controlled trial evaluating the efficacy of fractionated carbon dioxide therapy in postoperative lower extremity wound healing. This study, including analysis and submission for publication, will occur from September 2018 to November 2020. A cohort of 48 patients will be recruited. Eligibility criteria will include patients older than 18 years, those with a lower extremity wound as a result of Mohs Micrographic Surgery at Saint Louis University Dermatology Des Peres, and a postoperative wound greater than 5mm in diameter. Patients must be able to understand the informed consent, willing to come to the office for treatments and capable of following post-treatment instructions. Exclusion criteria will include pregnancy, immunosuppression, uncontrolled diabetes (defined as >7% A1c in the last 3 months), peripheral vascular disease, venous insufficiency, or no desire/unable to undergo laser therapy.

After informed consent is obtained, a screening visit will be performed on their Mohs surgery day and patient eligibility will be determined. Then, patients will be randomized 1:1 to a treatment or control group via computer software. One arm will receive carbon dioxide AFL immediately postoperatively on the wound base. The second arm, which will serve as control, will receive sham laser therapy. Both patients will be given identical postoperative wound care instructions, including vaseline applied to the wound, a piece of telfa to overlay the wound, and paper tape to secure the dressing. Additionally, patients will be advised to avoid baths and application of any other products to their wound. Patients will be given a diary to record observations about their postoperative wound and to note any adverse events.

Blinding

There will be one unblinded member of the team in this study which will be the clinician performing laser therapy or sham therapy, who will therefore not be involved in any data collection, but will be responsible for reporting any adverse events per IRB protocols at our institution. Other members of the research team member will be blinded to patient group assignment, and these members of the research team will collect data (see below) at subsequent visit. Additionally, patients will be blinded to treatment group. This will be achieved by having patients wear safety glasses which blind them and the wound site still anesthetized from the operation. Data collection will be done by a separate research team member who is blinded to the treatment groups.

Patient Visits and Data Collection

Patients will be seen at 4 separate visits. This will include the baseline visit and every 4 weeks to monitor safety and efficacy endpoints (4, 8 and 12 weeks post-operatively). The patient's initial visit will include preoperative screening for eligibility, informed consent procedure, and recording of past medical history and physical exam. Once the patient is deemed eligible, enrolled, and signed informed consent, they will be randomized to either carbon dioxide AFL therapy or sham laser therapy. After the patient undergoes Mohs surgery with the resultant ulcer (the defect that typically forms after Mohs), the patient will undergo either carbon dioxide laser versus sham laser therapy.

The investigators will look at the presence or absence of complete healing, wound temperature, a digital photograph, quality of life, and adverse events at each visit. Healing will be determined by one of the licensed research team members and will be defined by complete epithelialization in the absence of scab/eschar. Wound temperature will be recorded by non-invasive infrared thermographic camera. A digital photograph will be taken with a camera that has an attachment ensuring the same distance and angle at every visit. Quality of life will be determined by ED-5Q questionnaire. Adverse events will be recorded by eliciting an oral history and review of the patients diary. Adverse events will be recorded as presence of absence of specific outcomes. Outcomes that patients will be directly questioned about include: crusting (scaly or thickened scar), swelling, burning sensation, xerosis at treatment site, pruritus at treatment site, infection, bleeding, hypertrophic or keloid scarring, burns, or color changes at treatment site. These data points will be collected at every visit, and adjudicated by a member of the research team blinded to the treatment group. This member will be a licensed research team member.

Placebo treatment will consist of directing the laser system at the floor instead of the patient's wound site. The patients will be wearing safety glasses and will have their wound site still anesthetized from the operation therefore unaware if they are receiving the therapy. This group will serve as the control group to the treatment arm in the study.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Lower extremity wound as a result of Mohs Micrographic Surgery at Saint Louis University Dermatology Des Peres
* A postoperative wound greater than 5 mm in diameter
* Able to understand the informed consent, willing to come to the office for treatments and capable of following post-treatment instructions.

Exclusion Criteria:

* Pregnancy
* Breast feeding
* Immunosuppression
* Uncontrolled diabetes (defined as >7% A1c in the last 3 months)
* peripheral vascular disease
* venous insufficiency
* decompensated heart failure (NYHA class IV)
* peripheral neuropathy involving the treatment site
* active cancer at the time of study enrollment excluding curatively treated skin cancer
* Any underlying or current medical condition which, in the opinion of the Investigator, would interfere with the evaluation of the subject. or no desire/unable to undergo laser therapy.

Immunosuppression will be defined as patients with HIV, AIDS, who have received an organ transplant, allogeneic bone marrow transplant, or peripheral stem cell transplant, and any other patients taking chronic doses of systemic immunosuppressive medication within 6 months prior to randomization. Examples of immunosuppressive medications include Tacrolimus, Azathioprine, Prednisone, or Methotrexate.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rogers HW, Weinstock MA, Feldman SR, Coldiron BM. Incidence Estimate of Nonmelanoma Skin Cancer (Keratinocyte Carcinomas) in the U.S. Population, 2012. JAMA Dermatol. 2015 Oct;151(10):1081-6. doi: 10.1001/jamadermatol.2015.1187. PMID 25928283
- [Background] Subramaniam P, Olsen CM, Thompson BS, Whiteman DC, Neale RE; QSkin Sun and Health Study Investigators. Anatomical Distributions of Basal Cell Carcinoma and Squamous Cell Carcinoma in a Population-Based Study in Queensland, Australia. JAMA Dermatol. 2017 Feb 1;153(2):175-182. doi: 10.1001/jamadermatol.2016.4070. PMID 27892984
- [Background] Richmond-Sinclair NM, Pandeya N, Ware RS, Neale RE, Williams GM, van der Pols JC, Green AC. Incidence of basal cell carcinoma multiplicity and detailed anatomic distribution: longitudinal study of an Australian population. J Invest Dermatol. 2009 Feb;129(2):323-8. doi: 10.1038/jid.2008.234. Epub 2008 Jul 31. PMID 18668137
- [Background] Wei EX, Qureshi AA, Han J, Li TY, Cho E, Lin JY, Li WQ. Trends in the diagnosis and clinical features of melanoma in situ (MIS) in US men and women: A prospective, observational study. J Am Acad Dermatol. 2016 Oct;75(4):698-705. doi: 10.1016/j.jaad.2016.05.011. Epub 2016 Jul 16. PMID 27436155
- [Background] Honaker JS, Bordeaux JS, Tuttle MS. Retrospective Review of Risk Factors Predictive of Complications in Patients After Below the Knee Mohs Micrographic Surgery. Dermatol Surg. 2016 Apr;42(4):568-70. doi: 10.1097/DSS.0000000000000613. No abstract available. PMID 26949930
- [Background] Harlin SL, Harlin RD, Sherman TI, Rozsas CM, Shafqat MS, Meyers W. Using a structured, computer-administered questionnaire for evaluating health-related QOL with chronic lower extremity wounds. Ostomy Wound Manage. 2009 Sep 15;55(9):30-9. PMID 19797801
- [Background] Koupidis SA, Paraskevas KI, Stathopoulos V, Mikhailidis DP. Impact of lower extremity venous ulcers due to chronic venous insufficiency on quality of life. Open Cardiovasc Med J. 2008;2:105-9. doi: 10.2174/1874192400802010105. Epub 2008 Nov 28. PMID 19430523
- [Background] Demidova-Rice TN, Hamblin MR, Herman IM. Acute and impaired wound healing: pathophysiology and current methods for drug delivery, part 1: normal and chronic wounds: biology, causes, and approaches to care. Adv Skin Wound Care. 2012 Jul;25(7):304-14. doi: 10.1097/01.ASW.0000416006.55218.d0. PMID 22713781
- [Background] Singer AJ, Clark RA. Cutaneous wound healing. N Engl J Med. 1999 Sep 2;341(10):738-46. doi: 10.1056/NEJM199909023411006. No abstract available. PMID 10471461
- [Background] Persoon A, Heinen MM, van der Vleuten CJ, de Rooij MJ, van de Kerkhof PC, van Achterberg T. Leg ulcers: a review of their impact on daily life. J Clin Nurs. 2004 Mar;13(3):341-54. doi: 10.1046/j.1365-2702.2003.00859.x. PMID 15009337
- [Background] Herber OR, Schnepp W, Rieger MA. A systematic review on the impact of leg ulceration on patients' quality of life. Health Qual Life Outcomes. 2007 Jul 25;5:44. doi: 10.1186/1477-7525-5-44. PMID 17651490
- [Background] Lee SH, Zheng Z, Roh MR. Early postoperative treatment of surgical scars using a fractional carbon dioxide laser: a split-scar, evaluator-blinded study. Dermatol Surg. 2013 Aug;39(8):1190-6. doi: 10.1111/dsu.12228. Epub 2013 Apr 30. PMID 23631513
- [Background] Brandi C, Grimaldi L, Nisi G, Brafa A, Campa A, Calabro M, Campana M, D'Aniello C. The role of carbon dioxide therapy in the treatment of chronic wounds. In Vivo. 2010 Mar-Apr;24(2):223-6. PMID 20363999
- [Background] Schmitt L, Huth S, Amann PM, Marquardt Y, Heise R, Fietkau K, Huth L, Steiner T, Holzle F, Baron JM. Direct biological effects of fractional ultrapulsed CO2 laser irradiation on keratinocytes and fibroblasts in human organotypic full-thickness 3D skin models. Lasers Med Sci. 2018 May;33(4):765-772. doi: 10.1007/s10103-017-2409-1. Epub 2017 Dec 7. PMID 29218493
- [Background] Manstein D, Herron GS, Sink RK, Tanner H, Anderson RR. Fractional photothermolysis: a new concept for cutaneous remodeling using microscopic patterns of thermal injury. Lasers Surg Med. 2004;34(5):426-38. doi: 10.1002/lsm.20048. PMID 15216537
- [Background] Shumaker PR, Kwan JM, Badiavas EV, Waibel J, Davis S, Uebelhoer NS. Rapid healing of scar-associated chronic wounds after ablative fractional resurfacing. Arch Dermatol. 2012 Nov;148(11):1289-93. doi: 10.1001/2013.jamadermatol.256. PMID 23165834
- [Background] Phillips TJ, Morton LM, Uebelhoer NS, Dover JS. Ablative Fractional Carbon Dioxide Laser in the Treatment of Chronic, Posttraumatic, Lower-Extremity Ulcers in Elderly Patients. JAMA Dermatol. 2015 Aug;151(8):868-71. doi: 10.1001/jamadermatol.2015.0645. PMID 25946007

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fractional Carbon Dioxide Laser Intervention Group | Sham Laser Intervention Group
Started | 24 | 24
Completed | 23 | 21
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fractional Carbon Dioxide Laser Intervention Group | Sham Laser Intervention Group | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 18
  >=65 years | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (12) | 72 (12) | 71 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 38
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 22 | 24 | 46
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Completely Healed Lower Extremity Wounds
Description: Number of participants with completely healed lower extremity wounds by the end of the study (week 12). Complete wound healing is defined by reepithelization of the wound.
Time Frame: 12 weeks (enrollment time per subject)
Measure: Count of Participants; unit: Participants
Arm/Group | Fractional Carbon Dioxide Laser Intervention Group | Sham Laser Intervention Group
Number analyzed (Participants) | 23 | 21
Participants | 20 | 18

2. Primary Outcome: Number of Participants Who Experienced Adverse Events.
Description: Number of participants who experienced adverse events at any time point throughout the study.
Time Frame: 12 weeks (enrollment time per subject)
Measure: Count of Participants; unit: Participants
Arm/Group | Fractional Carbon Dioxide Laser Intervention Group | Sham Laser Intervention Group
Number analyzed (Participants) | 23 | 21
Participants | 4 | 2

3. Secondary Outcome: Quality of Life Measure EQ-5D-5L
Description: Score on the EQ-5D-5L. This is a quality of life questionnaire where higher scores equate to a better quality of life. The scale ranges from 100 ('the best imaginable health state' or 'the best health state you can imagine') to 0 ('the worst imaginable health state' or 'the worst health you can imagine').
Time Frame: 12 weeks (enrollment time per subject)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Fractional Carbon Dioxide Laser Intervention Group | Sham Laser Intervention Group
Number analyzed (Participants) | 23 | 21
scores on a scale | 90.7 (10.4) | 87.5 (10)

4. Secondary Outcome: Wound Temperature Associated With Carbon Dioxide Ablative Fractional Laser for Healing Postoperative Lower Extremity Wounds.
Description: Wound temperature will be recorded in degrees Celsius through an infrared camera.
Time Frame: 12 weeks (enrollment time per subject)
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Fractional Carbon Dioxide Laser Intervention Group | Sham Laser Intervention Group
Number analyzed (Participants) | 23 | 21
degrees Celsius | 32.41 (2.51) | 31.76 (1.98)

ADVERSE EVENTS:
Time Frame: Adverse events data was collected during the entire duration of the patient's enrollment in the study, which was until 12 weeks.
Description: Infection was diagnosed with a positive culture.
Arm/Group | Fractional Carbon Dioxide Laser Intervention Group | Sham Laser Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 4/24 | 2/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fractional Carbon Dioxide Laser Intervention Group (N=24) | Sham Laser Intervention Group (N=24)
Skin Infection (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/49/NCT03644849/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/49/NCT03644849/ICF_001.pdf